CLINICAL TRIAL: NCT04678310
Title: iLIVE Project: Live Well, Die Well. A Nested Volunteer Study
Brief Title: iLIVE Volunteer Study
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001538 iLIVE Volunteer
Record Dates: First submitted 2020-12-08; First posted 2020-12-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-07

CONDITIONS: Terminal Illness
Keywords: Dying; Palliative Care; Volunteers; End-of-Life-Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: A patient will be assessed as 'eligible' for participation in the iLIVE Volunteer Study if they have an advanced, incurable illness that is unlikely to be cured, and they have been assessed by their clinical team as being in the last month of life. If patients meet this criteria, they will be offered support from the hospital palliative and end of life care volunteer service (developed for this study). Patients who agree to support will be recruited to the 'Intervention Group'.
  Interventions: Other: Support from the hospital palliative and end of life care volunteer service (developed for this study).
- Case Control Comparison Group: If a patient is 'eligible' to receive support from the hospital palliative and end of life care volunteer service (see 'Intervention Group'), but declines involvement, they will be approached for inclusion in the study, as part of the 'Case Control Comparison' group for comparative analysis to assess the 'impact' of the volunteer service.

INTERVENTIONS:
Other: Support from the hospital palliative and end of life care volunteer service (developed for this study). — Hospital palliative and end of life care volunteer service: a volunteer service to provide support to patients dying in the hospital and their families. The volunteer service has been designed to provide presence and companionship to dying patients at the end of life, and their families.
  Groups: Intervention Group

SUMMARY:
The aim of this study is to develop and evaluate the implementation of an international volunteer training programme to support patients dying in the hospital setting and their families. It has the following objectives:

1. Explore the experience and perceptions of the international hospital palliative and end of life care volunteer programme, including care delivery, from the perspectives of:

   * Patients and their family members who receive the service
   * Volunteers who deliver the service
   * Health care professionals caring for patients who receive the service
2. Assess the implementation and impact of a hospital volunteer service for dying patients

DETAILED DESCRIPTION:
An excess of 5 million people die in the EU each year, with 77% of deaths resulting from chronic disease and illness. Of these 4 million deaths, many people will have died in pain or symptomatic distress, died alone, and/or died without structured health or social care for the patient and/or their family. Volunteer support represents an important and necessary community resource to enhance the experience of living at the end of life, and dying, however, a Cochrane review in 2015 concluded: "research is needed on the impact of training and support for palliative care volunteers on patients, their families, volunteers and palliative care services". Palliative care volunteer services are relatively uncommon and empirical evidence of the usefulness of such services in the hospital setting remains scarce.

An EU H2020 funded study, iLIVE, will address this concern. The iLIVE Volunteer Study, one of 8 workpackages within the iLIVE project, has developed an international hospital palliative care volunteer training programme, to support the implementation of palliative care volunteer services within five hospitals in five countries. The study will evaluate the implementation, use and experience of the iLIVE Volunteer Service across the five countries, embedded within the current iLIVE Cohort Study (ClinicalTrials.giv reference number: NCT04271085).

Aim/Rationale:

The aim of this study is to develop and evaluate the implementation of an international volunteer training programme to support patients dying in the hospital setting and their families.

Objectives:

1. Explore the experience and perceptions of the international hospital palliative and end of life care volunteer programme, including care delivery, from the perspectives of:

   1. Patients and their family members who receive the service
   2. Volunteers who deliver the service
   3. Health care professionals caring for patients who receive the service
2. Assess the implementation and impact of a hospital volunteer service for dying patients

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years old;
* The patient has already been recruited to the iLIVE Cohort Study (fulfilling the eligibility criteria);
* The physician or clinical team estimates the patient's life expectancy to be one month or less, based on a modified version of the 'Surprise Question' "Would you be surprised if this patient would die within one month?"
* The physician or clinical team agrees that the patient is eligible for involvement of the hospital palliative care volunteer service.

Exclusion Criteria:

* Patient is <18 years old;
* The patient has not already been recruited to the iLIVE Cohort Study and does not fulfil the eligibility criteria;
* The physician or clinical team does not estimate the patient's life expectancy to be one month or less, based on a modified version of the 'Surprise Question' "Would you be surprised if this patient would die within one month?"
* The physician or clinical team do not agree that the patient is eligible for involvement of the hospital palliative care volunteer service.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be any patient who is admitted to a participating hospital, and who meets the inclusion criteria for the study.
  All patients will have an advanced, incurable illness from which they will not be cured, and will have been assessed by their clinical team as being in the last month of life.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change over time, using the EuroQol Group 5-level EQ-5D version questionnaire (EQ-5D-5L). | Baseline (recruitment)
  The EQ-5D-5L is made up of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on 5 levels, using a 1-digit number: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems and 5 = extreme problems. The digits for the 5 dimensions are then combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled '100 = The best health you can imagine' and '0 = The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Assessment of change over time, using the EuroQol Group 5-level EQ-5D version questionnaire (EQ-5D-5L). | Follow-up 1 (7 days [+/- 2 days] following support from volunteer service)
  The EQ-5D-5L is made up of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on 5 levels, using a 1-digit number: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems and 5 = extreme problems. The digits for the 5 dimensions are then combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled '100 = The best health you can imagine' and '0 = The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Assessment of change over time, using the EuroQol Group 5-level EQ-5D version questionnaire (EQ-5D-5L). | Follow-up 2 (1 month following recruitment)
  The EQ-5D-5L is made up of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on 5 levels, using a 1-digit number: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems and 5 = extreme problems. The digits for the 5 dimensions are then combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled '100 = The best health you can imagine' and '0 = The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Assessment of change over time, using the Patient Capability Measure: ICECAP Supportive Care Measure (ICECAP-SCM). | Baseline (recruitment)
  ICECAP-SCM is a self-completion questionnaire developed to evaluate quality of life in palliative and supportive care.
  The ICECAP-SCM comprises 7 attributes: Having a say; Being with people who care about you; Physical suffering; Emotional suffering; Dignity; Being supported; Being prepared. Each dimension is scored on 4 levels ranging from: 4 = full capability; 1 = no capability. Higher scores indicate a better outcome.
Assessment of change over time, using the Patient Capability Measure: ICECAP Supportive Care Measure (ICECAP-SCM). | Follow-up 1 (7 days [+/- 2 days] following support from volunteer service)
  ICECAP-SCM is a self-completion questionnaire developed to evaluate quality of life in palliative and supportive care.
  The ICECAP-SCM comprises 7 attributes: Having a say; Being with people who care about you; Physical suffering; Emotional suffering; Dignity; Being supported; Being prepared. Each dimension is scored on 4 levels ranging from: 4 = full capability; 1 = no capability. Higher scores indicate a better outcome.
Assessment of change over time, using the Patient Capability Measure: ICECAP Supportive Care Measure (ICECAP-SCM). | Follow-up 2 (1 month following recruitment)
  ICECAP-SCM is a self-completion questionnaire developed to evaluate quality of life in palliative and supportive care.
  The ICECAP-SCM comprises 7 attributes: Having a say; Being with people who care about you; Physical suffering; Emotional suffering; Dignity; Being supported; Being prepared. Each dimension is scored on 4 levels ranging from: 4 = full capability; 1 = no capability. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Distress Thermometer (single measure questionnaire) | Follow-up 1 (7 days [+/- 2 days] following support from volunteer service); follow-up 2 (1 month following recruitment)
  The Distress Thermometer is a one-item self-report screening tool for measuring psychological distress in cancer patients. The scale is measured from 0 - 10, where a higher number indicates a better outcome: 0 = No Distress and 10 = Extreme Distress.

CONTACTS AND LOCATIONS:
Overall Officials: John E Ellershaw, Principal Investigator — University of Liverpool
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildiz B, van der Heide A, Bakan M, Iversen GS, Haugen DF, McGlinchey T, Smeding R, Ellershaw J, Fischer C, Simon J, Vibora-Martin E, Ruiz-Torreras I, Goossensen A; iLIVE consortium. Facilitators and barriers of implementing end-of-life care volunteering in a hospital in five European countries: the iLIVE study. BMC Palliat Care. 2024 Apr 2;23(1):88. doi: 10.1186/s12904-024-01423-5. PMID 38561727